CLINICAL TRIAL: NCT04407962
Title: PUSHME (Primary Care USage of Health Promoting Messages): A Text Message-based Intervention in Primary Care Patients With Hypertension: a Randomized Controlled Trial
Brief Title: Primary Care Usage of Health Promoting Messages
Acronym: PUSHME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-06361
Record Dates: First submitted 2020-05-25; First posted 2020-05-29 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Hypertension; Cardiovascular Risk Factor
Keywords: Hypertension; Text messaging; Primary Health Care; Health Promotion; Cardiovascular Risk Factor; Quality of Life
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMS group (Experimental): Participants in the intervention group will receive four semi-personalized messages per week in addition to their usual care according to the National Board of Health and Welfare guidelines for hypertension treatment.
  Interventions: Behavioral: SMS group
- Control group (No Intervention): The control group will receive usual care according to the National Board of Health and Welfare guidelines for hypertension treatment.

INTERVENTIONS:
Behavioral: SMS group — The experimental treatment will consist of health promoting text messages addressing metabolic risk factors associated with cardiovascular disorders in patients with hypertension. The text messages will be developed to support healthy life style changes i.e. regarding general cardiovascular health, tobacco use, physical activity and diet.
  Arms: SMS group

SUMMARY:
This project aims to investigate the use of e-health to assist health personnel in primary health care to carry out preventive measures of cardiovascular disease.The primary objective of the study is to examine the impact of lifestyle advices, administered through regularly sent SMS, on hypertension in a primary health care setting. The secondary objective is to evaluate changes in other cardiovascular risk factors and general health, e.g. tobacco use, obesity, blood lipids, HbA1c, self-rated health and health-related quality of life.

DETAILED DESCRIPTION:
This is a randomised controlled multi-centre study.The study will involve 400 patients from 9 primary health care centres located in four different regions in Sweden (Region Skåne, Region Kronoberg, Region Stockholm, Västra Götalandsregionen).

Patients in the intervention group will receive SMS messages aiming to remind, encourage and motivate patients to pursue healthy lifestyle changes. After baseline measurement, participants in the intervention group will receive four semi-personalized SMS messages per week for six months, in addition to their usual anti-hypertensive treatment. Each week, the participants will receive SMS from each of the following groups: A. Physical activity, B. Tobacco use, C. Dietary habits, and D. Cardiovascular health in general, except for non-smokers who, instead of the tobacco use-SMS, will get one extra randomly selected SMS.

Included patients that consent to take part in the study will be invited to their primary health care centre for a baseline visit. The following measurements will be assessed by a research assistant: blood pressure (in sitting position after 5 minutes rest; mean of two measurements in a standardized procedure with validated electronic BP devices), BMI and waist-hip circumference. Furthermore, the patients will complete a short questionnaire for evaluation of medical history, medication, tobacco and alcohol use, physical activity level, self-rated health and health-related quality of life. Blood samples for HbA1c and cholesterol will be drawn. Randomization will be performed after completion of baseline assessments and questionnaires. A follow up control will be performed after 6 months with the same assessments as at the baseline visit.

The primary endpoint is change inblood pressure (mmHg). Secondary endpoints are changes in Cholesterol (total cholesterol, high-density lipoprotein [HDL], low-density lipoprotein [LDL]) (mmol/l), Tobacco and alcohol use, BMI (kg/m2), waist circumference, HbA1c (mmol/mol), Self-rated health (five-graded Likert scale), Health related quality of life, as measured by EQ5D-5L, Self-reported physical activity.

The power analysis indicates a sample size of 189 patients in each arm. The calculation is based on an assumed statistical power of 80%, a two-sided test, using a significant level of 5% with a difference of 4 mm Hg between the groups, a standard deviation of 13 mm Hg and a drop out rate of 15%. Data will be analyzed according to the intention-to-treat principle. Differences in mean change of endpoints between intervention and control groups will be calculated by ANCOVA, with baseline values as covariates. Correlation between behavioral change (smoke cessation,increased level of physical activity) and behavioral predictors will be analyzed with logistic regression analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with hypertension (defined by the International classification of disease Manual ICD-10, diagnose code I10.9)
2. 40-85 years
3. Patient must own a smart mobile phone

Exclusion Criteria:

1. Blood pressure at baseline visit ≥180/110 mmHg or systolic blood pressure<120 mmHg
2. Serious illness with short life expectancy (<1year)
3. Predicted inability to comply with the study protocol e.g. language difficulties, interpreter needs, serious cognitive impairment
4. Pregnancy

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | six months
  Measured by automated devices (mmHg)

SECONDARY OUTCOMES:
Changes in cholesterol | six months
  Measured by blood test, total cholesterol (mmol/l)
Changes in high-density lipoprotein [HDL] | six months
  Measured by blood test, high-density lipoprotein [HDL] (mmol/l)
Changes in low-density lipoprotein [LDL] | six months
  Measured by blood test, low-density lipoprotein [LDL] (mmol/l)
Changes in tobacco use | six months
  self-reported. Do you smoke?: 1. Yes, 2. No, 3. Previous smoker. Any changes during study period will be registered.
Changes in Blood glucose | six months
  HbA1c
Changes in self-rated health | six months
  five-graded Likert scale from excellent to poor. The question posed is; in general, would you say that you health is excellent, very good, good, fair, or poor?
Changes in self rated quality of life | six months
  EQ5D-5L (EuroQol 5 dimentions).The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.
Changes in level of physical activity | six months
  self-reported physical activity: How much time do you spend during a typical week doing physical exercise, which will make you feel short of breath, such as running, fitness calsses, ball sports? 1. No time, 2. 0-29 min, 3. 30-59 min, 4. 60-120 min, 5.>120 minHow much time do you spend during a typical week doing everyday exercise, such as walking, cycling, gardening? Adding together all the time (at least 10 minutes at the time) 1. No time, 2. 0-29 min, 3. 30-59 min, 4. 60-119 min, 5. 2-3 h, 6. >3-5 h, 7. >5 h
Changes in alcohol use | six months
  self-reported. Do you drink alcohole? (wine, beer or spirits) See explanation of the term "standard glass of alcohole" 1. No, or <1 glass/w, 2. 1-4 g/w, 3. 5-8 g/w, 4. 9-12 g/w, 5. 13-19 g/w, 6. >20g/w

CONTACTS AND LOCATIONS:
Locations (9):
- Sweden (9):
  - Bokskogens Health Care Center, Bara
  - Laröds Health Care Center, Helsingborg
  - Vårdcentralen Delfinen, Höganäs
  - Vårdcentralen Nötkärnan, Kållered
  - Nöbbelövs Health Care Center, Lund
  - Rävlanda vårdcentral, Rävlanda
  - Närhälsan Tidaholm, Tidaholm
  - Skärvet Health Care Center, Vaxjo
  - Hovshaga Health Care Center, Vaxjo

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data will be approved by a review committee for this purpose.

REFERENCES:
- [Background] NCD Risk Factor Collaboration (NCD-RisC). Worldwide trends in blood pressure from 1975 to 2015: a pooled analysis of 1479 population-based measurement studies with 19.1 million participants. Lancet. 2017 Jan 7;389(10064):37-55. doi: 10.1016/S0140-6736(16)31919-5. Epub 2016 Nov 16. PMID 27863813
- [Background] GBD 2016 Risk Factors Collaborators. Global, regional, and national comparative risk assessment of 84 behavioural, environmental and occupational, and metabolic risks or clusters of risks, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1345-1422. doi: 10.1016/S0140-6736(17)32366-8. PMID 28919119
- [Background] Schillaci G, Pirro M, Vaudo G, Gemelli F, Marchesi S, Porcellati C, Mannarino E. Prognostic value of the metabolic syndrome in essential hypertension. J Am Coll Cardiol. 2004 May 19;43(10):1817-22. doi: 10.1016/j.jacc.2003.12.049. PMID 15145106
- [Background] Alberti KG, Eckel RH, Grundy SM, Zimmet PZ, Cleeman JI, Donato KA, Fruchart JC, James WP, Loria CM, Smith SC Jr; International Diabetes Federation Task Force on Epidemiology and Prevention; Hational Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; International Association for the Study of Obesity. Harmonizing the metabolic syndrome: a joint interim statement of the International Diabetes Federation Task Force on Epidemiology and Prevention; National Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; and International Association for the Study of Obesity. Circulation. 2009 Oct 20;120(16):1640-5. doi: 10.1161/CIRCULATIONAHA.109.192644. Epub 2009 Oct 5. PMID 19805654
- [Background] Grundy SM. Metabolic syndrome update. Trends Cardiovasc Med. 2016 May;26(4):364-73. doi: 10.1016/j.tcm.2015.10.004. Epub 2015 Oct 31. PMID 26654259
- [Background] Lindblad U, Ek J, Eckner J, Larsson CA, Shan G, Rastam L. Prevalence, awareness, treatment, and control of hypertension: rule of thirds in the Skaraborg project. Scand J Prim Health Care. 2012 Jun;30(2):88-94. doi: 10.3109/02813432.2012.684207. PMID 22643153
- [Background] Cottrell E, Chambers R, O'Connell P. Using simple telehealth in primary care to reduce blood pressure: a service evaluation. BMJ Open. 2012 Oct 31;2(6):e001391. doi: 10.1136/bmjopen-2012-001391. Print 2012. PMID 23117563
- [Background] Arambepola C, Ricci-Cabello I, Manikavasagam P, Roberts N, French DP, Farmer A. The Impact of Automated Brief Messages Promoting Lifestyle Changes Delivered Via Mobile Devices to People with Type 2 Diabetes: A Systematic Literature Review and Meta-Analysis of Controlled Trials. J Med Internet Res. 2016 Apr 19;18(4):e86. doi: 10.2196/jmir.5425. PMID 27095386
- [Background] Mussener U, Bendtsen M, Karlsson N, White IR, McCambridge J, Bendtsen P. Effectiveness of Short Message Service Text-Based Smoking Cessation Intervention Among University Students: A Randomized Clinical Trial. JAMA Intern Med. 2016 Mar;176(3):321-8. doi: 10.1001/jamainternmed.2015.8260. PMID 26903176
- [Background] Bengtsson U, Kjellgren K, Hallberg I, Lindwall M, Taft C. Improved Blood Pressure Control Using an Interactive Mobile Phone Support System. J Clin Hypertens (Greenwich). 2016 Feb;18(2):101-8. doi: 10.1111/jch.12682. Epub 2015 Oct 12. PMID 26456490
- [Background] Chow CK, Redfern J, Hillis GS, Thakkar J, Santo K, Hackett ML, Jan S, Graves N, de Keizer L, Barry T, Bompoint S, Stepien S, Whittaker R, Rodgers A, Thiagalingam A. Effect of Lifestyle-Focused Text Messaging on Risk Factor Modification in Patients With Coronary Heart Disease: A Randomized Clinical Trial. JAMA. 2015 Sep 22-29;314(12):1255-63. doi: 10.1001/jama.2015.10945. PMID 26393848
- [Background] Margolis KL, Asche SE, Bergdall AR, Dehmer SP, Maciosek MV, Nyboer RA, O'Connor PJ, Pawloski PA, Sperl-Hillen JM, Trower NK, Tucker AD, Green BB. A Successful Multifaceted Trial to Improve Hypertension Control in Primary Care: Why Did it Work? J Gen Intern Med. 2015 Nov;30(11):1665-72. doi: 10.1007/s11606-015-3355-x. PMID 25952653
- [Background] Godin G, Kok G. The theory of planned behavior: a review of its applications to health-related behaviors. Am J Health Promot. 1996 Nov-Dec;11(2):87-98. doi: 10.4278/0890-1171-11.2.87. PMID 10163601
- [Background] Johnston DW, Johnston M, Pollard B, Kinmonth AL, Mant D. Motivation is not enough: prediction of risk behavior following diagnosis of coronary heart disease from the theory of planned behavior. Health Psychol. 2004 Sep;23(5):533-8. doi: 10.1037/0278-6133.23.5.533. PMID 15367073
- [Background] Palmeira AL, Teixeira PJ, Branco TL, Martins SS, Minderico CS, Barata JT, Serpa SO, Sardinha LB. Predicting short-term weight loss using four leading health behavior change theories. Int J Behav Nutr Phys Act. 2007 Apr 20;4:14. doi: 10.1186/1479-5868-4-14. PMID 17448248
- [Background] Owen N, Sugiyama T, Eakin EE, Gardiner PA, Tremblay MS, Sallis JF. Adults' sedentary behavior determinants and interventions. Am J Prev Med. 2011 Aug;41(2):189-96. doi: 10.1016/j.amepre.2011.05.013. PMID 21767727
- [Derived] Brodin N, Wolff M, Borgstrom Bolmsjo B, Milos Nymberg V, Nymberg P, Calling S. Factors associated with blood pressure control in Swedish primary care patients with hypertension: a cross-sectional study. Scand J Prim Health Care. 2025 Jun 30:1-9. doi: 10.1080/02813432.2025.2524366. Online ahead of print. PMID 40583484
- [Derived] Borgstrom Bolmsjo B, Bredfelt J, Calling S, Glock H, Nymberg VM, Bengtsson Bostrom K, Jakobsson U, Nymberg P, Pallon J, Roost M, Wolff M. Health-promoting text messages to patients with hypertension-A randomized controlled trial in Swedish primary healthcare. PLoS One. 2025 Feb 12;20(2):e0314868. doi: 10.1371/journal.pone.0314868. eCollection 2025. PMID 39937817